CLINICAL TRIAL: NCT05350124
Title: The Effect of Vitamin C and E Therapy on Restless Leg Syndrome in Patients With End Stage Renal Disease on Haemodialysis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Siraj Omar Wali, Head of Sleep Medicine and research center, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VIT.C&E RLS on HM
Record Dates: First submitted 2022-03-17; First posted 2022-04-27 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Restless Legs Syndrome; End Stage Renal Disease
MeSH Terms: conditions — Restless Legs Syndrome; Kidney Failure, Chronic | interventions — Ascorbic Acid; Tocopherols; Vitamin E

STUDY DESIGN:
Intervention Model Description: randomization into four groups, each group will include 40 patients. A. Group 1: Will receive vitamin C (200 mg) tablet and vitamin E (a-tocopherol) (400 mg) capsule every day for 12 weeks. B. Group 2: Will receive vitamin E (400 mg) capsule and placebo every day for 12 weeks.
  C. Group 3: Will receive vitamin C (200 mg) tablet and placebo every day for 12 weeks. D. Group 4: Will receive two placebo every day for 12 weeks. Of note, the personal responsible for randomization will not be involved in the trial.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Vitamin C (200 mg) capsule, and vitamin E (400 IU) capsule every day for 12 weeks.
  Interventions: Drug: Ascorbic acid; Drug: Tocopherol
- Group 2 (Experimental): Vitamin C (200 mg) capsule, and placebo every day for 12 weeks.
  Interventions: Drug: Ascorbic acid; Drug: Placebo capsule
- Group 3 (Experimental): Vitamin E (400 IU) capsule, and placebo every day for 12 weeks.
  Interventions: Drug: Tocopherol; Drug: Placebo capsule
- Group 4 (Experimental): Placebo capsule (2 pills) every day for 12 weeks.
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: Ascorbic acid — vitamin C (200 mg) capsule
  Other Names: Vitamin C
  Arms: Group 1; Group 2
Drug: Tocopherol — vitamin E (400 IU) capsule
  Other Names: Vitamin E
  Arms: Group 1; Group 3
Drug: Placebo capsule — Placebo one pill only
  Other Names: Inactive substance
  Arms: Group 2; Group 3
Drug: Placebo capsule — Placebo two pills only
  Other Names: Inactive substance
  Arms: Group 4

SUMMARY:
This study aims to measure the effectiveness of vitamins C and E on relieving RLS symptoms in end stage renal disease patients on HD

DETAILED DESCRIPTION:
double-blind placebo-controlled trial of 12 weeks duration on end stage renal disease (ESRD) patients on HD with RLS.

All ESRD patients on HD will be screened clinically for RLS using the five diagnostic criteria of IRLSSG by trained physicians. then the Quastioniare will be filled and inclusion and exclusion criteria be checked sleep study must be done.

Each patient will then undergo a full sleep study using level 2 polysomnography at home. Periodic leg movements with sleep (PLMs) index and leg movements index (LM) before sleep onset will be recorded as well as other variables

Then Subjects will then be randomly assigned by blocked randomization into four groups, each group will include 40 patients. A. Group 1: Will receive vitamin C (200 mg) tablet and vitamin E (a-tocopherol) (400 mg) capsule every day for 12 weeks. B. Group 2: Will receive vitamin E (400 mg) capsule and placebo every day for 12 weeks.

C. Group 3: Will receive vitamin C (200 mg) tablet and placebo every day for 12 weeks. D. Group 4: Will receive two placebo every day for 12 weeks. Of note, the personal responsible for randomization will not be involved in the trial.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease patients on hemodialysis who met the five diagnostic criteria of RLS.

Exclusion Criteria:

* Secondary causes of RLS Medications (list included in section C below) iron deficiency or peripheral neuropathy

Presence of RLS-mimicking disorders:

1. Arthritis
2. Deep venous thrombosis
3. Varicose veins or venous insufficiency
4. Habitual foot tapping

Patients receiving medications that could trigger RLS:

1. Anticonvulsants, e.g., new use of anticonvulsant drugs within6 months of screening. A stable regimen of anticonvulsants was allowed.
2. Antipsychotics (haloperidol or phenothiazine derivatives)
3. Antidepressants (selective serotonin reuptake inhibitors or tricyclic antidepressants)
4. Antimanic (lithium)

Patients on medications or with conditions that may interfere with vitamin C & E absorption:

1. Celiac disease
2. Crohn's disease
3. Chronic pancreatitis
4. Cystic fibrosis
5. Weight-reduction drugs
6. Chemotherapy and radiotherapy

Patients with contraindications for vitamin C & E supplements:

1. Blood disorders, e.g., thalassemia, G6PD, sickle cell disease and hemochromatosis
2. Other conditions like diabetic patients, oxalate nephropathy, nephrolithiasis and vitamin E or C allergy
3. Unstable vital signs
4. Retinal eye disease
5. Cancers
6. Liver disease
7. Vitamin K deficiency

For women only:

1. Pregnancy (positive pregnancy test at screening)
2. Currently breastfeeding
3. Use of oral contraceptives or start of menopausal hormone therapy within 3 months of baseline

History of vitamin E or C intolerance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
International Restless Legs Syndrome Study Group (IRLSSG) diagnostic criteria | in screening
  The IRLSSG is a validated and reliable questionnaire. Well-trained physicians will aid patients in completing this questionnaire and perform clinical examination. It consists of five yes/no questions, subjects will be considered to have RLS if their answers are yes to all five questions
Stop Bang | in screening
  The STOP-Bang questionnaire includes the four questions used in the STOP questionnaire plus four additional demographic queries, for a total of eight dichotomous (yes/no) questions related to the clinical features of sleep apnea (snoring, tiredness, observed apnea, high blood pressure, BMI, age, neck circumference and male gender). For each question, answering "yes" scores 1, a "no" response scores 0, and the total score ranges from 0 to 8.
  Low Risk: Yes to 0 - 2 questions
  Intermediate Risk: Yes to 3 - 4 questions
  High Risk: Yes to 5 - 8 questions
  or Yes to 2 or more of 4 STOP questions + male gender
  or Yes to 2 or more of 4 STOP questions + BMI > 35kg/m2
  or Yes to 2 or more of 4 STOP questions + neck circumference 16 inches / 40cm
Hemoglobin | in screening
  Participants with normal levels between 12 - 15 g/dl Participants with levels below 12 or above 15 will be considered abnormal
Changes in The International Restless Leg Syndrome Study Group (IRLSSG) rating scale for restless legs syndrome | base line then once weekly for 12 weeks
  That consists of 10 questions scored from 0-4 with a total score ranging from 0-40 in which RLS severity is directly proportional to the total score. Meaning the higher the score, the worse and severe the symptoms.
Epworth sleepiness scale (ESS) | base line then once every 4 weeks for 12 weeks
  It is a self-administered questionnaire that measures the severity of excessive daytime sleepiness (EDS) containing 8 questions, each question is given a score from 0 to 3 with a total score of 0-24. A score above 10 is considered abnormal i.e. in keeping with EDS
Medical Outcomes Study Sleep Scale (MOS) | base line then once every 4 weeks for 12 weeks
  A 12-item scale that investigates six factors including; sleep initiation, respiratory problems, maintenance, perceived adequacy and somnolence. With higher score indicating higher sleep disturbance.
Suggested Immobilization Test (SIT) | base line then once every 4 weeks for 12 weeks
  prior to the sleep recording. at 45-degree angle with their legs outstretched. avoid moving voluntarily for the entire duration of the test. Surface EMG from the left and right anterior tibialis muscles is used to quantify leg movements. The latter are scored according to the criteria (movements lasting between 0.5 and 10 seconds, separated by intervals of 4 to 90 seconds and arising in series of at least 4 consecutive movements). The SIT periodic leg movements index represents the number of periodic leg movements per hour of immobility. Patients report severity of leg discomfort on a visual analogue scale (VAS) ranging from 0 (no discomfort) to 100 (extreme discomfort) every 10 minutes during the SIT. The mean leg discomfort score is assessed using the average of the 7 values, as well as the discomfort severity at the end of the test (time 60 minutes), the maximum leg discomfort during the test, and the variation between the lowest and the highest values recorded during the test
Restless Leg Syndrome (RLS) Symptoms Diary | base line then daily for the last 2 weeks
  The (RLS) Symptom Diary is a convenient tool to record information on your daily (RLS) symptoms, their duration, sleep patterns and possible triggers such as nicotine, alcohol or caffeine. to identify what influences, triggers or worsen the (RLS) symptoms
Polysomnography | base line then once every 4 weeks for 12 weeks
  Polysomnography (SOMNO Medics Plus; SOMNOmedics, Randersacker, Germany) consists of continuous recordings from surface leads for electroencephalography (EEG), electrooculography, electromyography (submental and bilateral anterior tibialis muscles), electrocardiography, nasal pressure, nasal and oral airflow (thermocouple), chest and abdominal impedance belts for respiratory muscle efforts, pulse oximetry for oxygen saturation and pulse rate, a tracheal microphone for snoring, and body position sensors for sleep position. PSG records are scored manually according to the American Academy of Sleep Medicine (AASM) 2020 scoring
Hemoglobin A1C | In screening
  Participants will be considered normal if the level is within 4.2 - 6.3 % Participants with a level higher than 6.3% will be considered abnormal
Vitamin D | In screening
  Participants will be considered normal if the level is within 75 - 250 nmol/L Participants will be considered abnormal if the level is less than 75 or higher than 250 nmol/L
Serum Iron | In screening
  Participants will be considered normal if the level is within 6 - 26 umol/L
Total Iron Binding Capacity | In screening
  Participants will be considered normal if the level is within 25 - 92 umol/L
Ferritin | In screening
  Participants will be considered normal if the level is within 13-150 ng/ml
Magnesium | In screening
  Participants will be considered normal if the level is within 1.7 - 2.2 mg/dL

IPD SHARING:
Plan to Share IPD: No